CLINICAL TRIAL: NCT00368901
Title: A Multicenter Study Using Once Every Other Week Subcutaneous Administration of Aranesp™ (Darbepoetin Alfa) and Iron Guided Algorithms to Treat Subjects With Anemia of Chronic Renal Insufficiency (CRI)
Brief Title: STAAR-2 Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20010215
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Kidney Disease; Chronic Renal Insufficiency; Kidney Disease; Pre-dialysis; Pre-ESRD
Keywords: Aranesp; Anemia; Kidney Disease; Hemoglobin; darbepoetin alfa; QoL
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Anemia | interventions — Darbepoetin alfa

ARMS (1):
- Single arm (Experimental): Every other week dosing of Aranesp SC
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Aranesp administered every other week SC titrated to not exceed Hb 12 g/dL
  Other Names: Aranesp

SUMMARY:
To assess the effect of Aranesp on the hemoglobin (Hgb) of CRI subjects who are recombinant human erythropoietin (rHuEPO)-naïve or converting from rHuEPO therapy.

DETAILED DESCRIPTION:
To assess the effect of Aranesp_ on the hemoglobin (Hgb) of CRI subjects who are recombinant human erythropoietin (rHuEPO)-naïve or converting from rHuEPO therapy. To assess the association between subject self-reported health-related quality of life (HRQoL) as it relates to Hgb concentration and glomerular filtration rate (GFR) in subjects who were rHuEPO-naïve prior to study enrollment. To characterize the health-related resource utilization of subjects with CRI. To characterize the subject satisfaction with Aranesp_ compared to previous rHuEPO therapy. To characterize iron treatment in subjects with CRI. To assess the safety profile of Aranesp_ therapy in subjects with CRI

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* diagnosis of CRI and not receiving dialysis therapy (must be predialysis)
* measured or estimated (using the Cockcroft-Gault formula) creatinine clearance (CrCl) of ≤ 70 mL/min, or GFR ≤ 60 mL/min (using the MDRD formula):
* Cockcroft-Gault formula: CrCl = (140 minus age in years) x (body weight in kg) serum creatinine (mg/dL) x 72.0 For women, the value will be multiplied by 0.85
* MDRD formula: GFR = 170 x [SCr]-0.999 x [Age]-0.167 x [0.762 if subject is female] x [1.180 if subject is black] x [sun] -0.170SAlb]-0.318
* mean Hgb < 11 g/dL during the screening/baseline period (if subject is not already receiving rHuEPO therapy)
* for subjects currently receiving rHuEPO therapy, the subject must have: a stable rHuEPO dose for the past month; and a rHuEPO frequency of once weekly.
* white blood cell and platelet counts within normal limits
* serum vitamin B12 and folate levels above the lower limit of normal range
* transferrin saturation (TSAT) ≥ 20% during the screening period
* availability for follow-up assessments
* subject must be able to comprehend and be willing to, or have legally accepted representative, give written informed consent for participation in the study

Exclusion Criteria:

* scheduled to initiate dialysis
* uncontrolled hypertension (diastolic blood pressure > 105 mm Hg or systolic blood pressure of > 180 mm Hg during the screening/baseline period on two separate measurements)
* clinically unstable in the judgment of the investigator (eg, subject is in the intensive care unit, immediately post-myocardial infarction, etc)
* scheduled to receive a living donor kidney transplant
* treatment of grand mal epilepsy within the past 6 months
* moderate to severe congestive heart failure (NYHA class III or IV)
* clinical evidence of severe secondary hyperparathyroidism (parathyroid hormone level > 1500 pg/mL)
* severe active chronic inflammatory process (eg, ulcerative colitis, peptic ulcer disease, rheumatoid arthritis, etc)
* currently receiving antibiotic therapy for systemic infection (enrollment may be postponed until the course of antibiotics has ended)
* known aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 3 times the upper limit of the normal range on more than one occasion within three months prior to screening
* known positive HIV antibody or hepatitis B surface antigen
* clinical evidence of current malignancy and/or receiving chemotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia
* active bleeding or RBC transfusion within eight weeks of enrollment
* androgen therapy within four weeks before enrollment
* known hematologic disease (eg, sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma; hemolytic anemia, etc)
* any condition that is likely to affect subject compliance
* currently or previously (within 30 days) enrolled in investigational device or drug trial(s) or receiving investigational agent(s)
* the exception to this is if the subject was enrolled in another Aranesp™ or rHuEPO protocol
* pregnant or breast feeding women (women of child-bearing potential must be using contraceptive precautions)
* women planning to have a child during the study period
* known hypersensitivity to the active substance or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2002-01; Primary Completion 2004-03 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Mean hemoglobin during the evaluation period | 52 weeks

SECONDARY OUTCOMES:
Change in hemoglobin throughout the study | 52 weeks
HRQoL scores of rHuEPO-naïve subjects measured at baseline, week 12, week 24, and end of study | 52 weeks
Health-related resource utilization, measured every 4 weeks, throughout the study | 52 weeks
Patient satisfaction scores of subjects previously on rHuEPO therapy, measured at baseline and week 12 | 12 weeks
Iron requirement (dose, frequency, and route) of subjects during the study | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Abu-Alfa AK, Sloan L, Charytan C, Sekkarie M, Scarlata D, Globe D, Audhya P. The association of darbepoetin alfa with hemoglobin and health-related quality of life in patients with chronic kidney disease not receiving dialysis. Curr Med Res Opin. 2008 Apr;24(4):1091-100. doi: 10.1185/030079908x280653. Epub 2008 Mar 6. PMID 18328118
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com